CLINICAL TRIAL: NCT04105231
Title: Cannabidiol for Treatment of Non-affective Psychosis and Cannabis Use
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lone Baandrup (Other)
Collaborators: Danish Center for Sleep Medicine (Other); Copenhagen University Hospital, Denmark (Other); Glostrup University Hospital, Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Lone Baandrup, Head of Clinic, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-P; 2018-004893-84 (EudraCT Number)
Record Dates: First submitted 2019-09-22; First posted 2019-09-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dual Diagnosis
Keywords: psychosis; cannabis; clinical trial
MeSH Terms: conditions — Psychotic Disorders; Marijuana Abuse | interventions — Cannabidiol; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Cannabidiol (Epidiolex®) (oral suspension)100 mg/ml dosed as 3 ml in the morning for 4 days, then increased to 3 ml in the morning and 3 ml in the evening, equivalent to CBD 300 mg BID, with a total treatment duration of 7 weeks.
  AND Risperione placebo, encapsulated tablet.
  Interventions: Drug: Cannabidiol
- Risperidone (Active Comparator): Risperidone (encapsulated tablet) dosed as 2 mg in the morning for 4 days, then increased with 2 mg in the morning and 2 mg in the evening, with a total treatment duration of 7 weeks
  AND Cannabidiol placebo, oral suspension
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol oral suspension
  Other Names: Epidiolex
  Arms: Cannabidiol
Drug: Risperidone — Risperidone, encapsulated tablet.
  Other Names: Risperidon
  Arms: Risperidone

SUMMARY:
This trial examines the efficacy of cannabidiol (CBD) versus risperidone for treatment of psychosis in patients with non affective-psychosis and lifetime use of cannabis.

DETAILED DESCRIPTION:
People with psychosis and comorbid cannabis use are particularly difficult to treat because cannabis use worsens psychotic symptoms and increases the risk that a first-episode psychosis will progress to schizophrenia. It is the THC (tetrahydrocannabinol) content in cannabis that aggravates psychotic symptoms whereas the CBD content has potential therapeutic effects. This trial investigates treatment with CBD (without THC) versus risperidone (an antipsychotic agent) in people with psychosis and lifetime use of cannabis. We hypothesize that CBD will ameliorate psychotic symptoms and reduce the frequency of cannabis use to a larger extent than risperidone. Sleep disturbances are often a limiting factor in the treatment of psychosis, and it is also examined how CBD affects objective and subjective sleep quality as well as circadian rest-activity cycles. Based on previous studies investigating CBD as monotherapy in patients with schizophrenia, it is expected that CBD will be associated with fewer adverse events than risperidone.

ELIGIBILITY:
Inclusion criteria:

* ICD-10 diagnosis of schizophrenia (DF20.X), paranoid psychosis (DF22.X), acute/intermittent psychotic disorder (DF23.X), schizoaffective psychosis (DF25.X), other/not specified nonorganic psychotic disorder (DF28/DF29), or cannabis induced psychotic disorder (DF12.5)
* PANSS ≥ 60 and score of ≥ 4 on ≥ 2 PANSS-Positive subscale items: Delusions (P1), conceptual disorganization (P2), hallucinatory behaviour (P3), grandiosity (P5), suspiciousness (P6)
* Lifetime cannabis use
* Age 18-45 years
* Female patients of childbearing potential need to utilize a proper method of contraception

Exclusion criteria:

* Treatment resistance as defined by treatment (ever) with clozapine
* Dependence syndrome of alcohol or psychoactive substances other than cannabis (DF1X.2 other than DF12.2)
* Psychotic disorder induced by alcohol or psychoactive substances other than cannabis (DF1X.5 other than DF12.5)
* Treatment with a long-acting injectable antipsychotic within the past month (or corresponding to the usual interval between two injections)
* Treatment with an oral antipsychotic within the past 7 days
* Use of self-administered CBD products during the trial
* Patients involuntarily admitted
* Pregnancy or lactation
* Severe physical illness that might influence the ability to comply with the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Psychotic symptoms | 7 weeks follow-up
  Positive and Negative Syndrome Scale (PANSS) positive subscale, range 7-49. A measure of symptom severity. Higher values are worse.

SECONDARY OUTCOMES:
Cannabis cessation (no use of cannabis within the past two weeks) (for current cannabis users at baseline) | 7 weeks follow-up
  Timeline follow back method
Cannabis use by self-reported days of cannabis use per week, since last study visit. | 7 weeks follow-up
  Timeline follow back method
Amount of cannabis use per day, self-reported, since last study visit. | 7 weeks follow-up
  PSYSCAN cannabis questionnaire# 6-8
Response | 7 weeks follow-up
  Response defined by PANSS total 25 percentile changes
Remission | 7 weeks follow-up
  Symptomatic remission is defined according to the Andreasen et al remission criteria. The criteria define symptomatic remission as a rating of no more than mild in four core positive and four core negative symptoms on the Positive and Negative Syndrome Scale (P1, P2 P3, N1, N4, N6, G5, G9,) that is sustained for ≥6 months. Because of the duration of this study, the requirement of 6 month will not be considered.
Global illness severity | 7 weeks follow-up
  Global illness severity is assessed with the Clinical Global Impression Scale (CGI). We will use the severity (CGI-S) at baseline and improvement (CGI-I) scores of the CGI at the following visits. Response will be defined as much improved or better on the CGI-I. The main item 'severity of illness' is measured on a 7-point Likert scale (from 1 'normal, not at all ill' to 7 'among the most extremely ill patients').
Psychosocial functioning | 7 weeks follow-up
  Personal and Social Performance Scale (PSP). Higher is better, range 1-100.
Neurocognitive functioning | 7 weeks follow-up
  Brief Assessment of Cognition in Schizophrenia (BACS). Neurocognitive Test Battery. One composite score and six subscales.
Subjective well-being | 7 weeks follow-up
  Subjective Well-being under Neuroleptics Scale (SWN). A measure of health-related quality of life.
Circadian rest-activity cycle | 7 weeks follow-up
  Actigraphy. A wrist-worne device that measures kinetic energy.
Subjective sleep quality | 7 weeks follow-up
  Pittsburgh Sleep Quality Index (PSQI). One total score, seven subscales.
Objective sleep evaluation | 7 weeks follow-up
  Polysomnography (PSG). A measure of objective sleep variables
Metabolomics | 7 weeks follow-up
  Markers for cannabinoids, dopamine and serotonin and their precursors and metabolites in the blood

OTHER OUTCOMES:
Adverse events (AEs), discontinuation due to AEs, and serious adverse events (SAEs) | From baseline to 2 weeks after end of treatment
  Self-report
Extrapyramidal and other side effects | 7 weeks follow-up
  Udvalget for Kliniske Undersoegelser (UKU) short version A clinician-rated scale to assess antipsychotic side effects

CONTACTS AND LOCATIONS:
Overall Officials: Lone Baandrup, MD, PhD, Principal Investigator — Mental Health Services Capital Region in Denmark
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available. In addition, the study protocol will be available. Data will be available after publication of planned primary and secondary analyses. There will be no end date for availability of data. Individual participant data will be available for meta-analysis. Proposals should be directed to: lone.baandrup@regionh.dk. To gain access, data requestors will need to sign a data access agreement.
Time Frame: Data will be available after publication of planned primary and secondary analyses. No end date.
Access Criteria: Proposals should be directed to: lone.baandrup@regionh.dk. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Rasmussen JO, Jennum P, Linnet K, Glenthoj BY, Baandrup L. Cannabidiol versus risperidone for treatment of recent-onset psychosis with comorbid cannabis use: study protocol for a randomized controlled clinical trial. BMC Psychiatry. 2021 Aug 14;21(1):404. doi: 10.1186/s12888-021-03395-9. PMID 34391393

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT04105231/SAP_000.pdf